CLINICAL TRIAL: NCT05868772
Title: What is the Efficiency When Comparing Active Sentry at Low IOP vs Ozil at High IOP?
Status: Completed | Type: Observational
Sponsor: Cataract and Laser Institute of Southern Oregon (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: JS-23-01
Record Dates: First submitted 2023-05-03; First posted 2023-05-22 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Active Sentry Handpiece: At low IOP settings
  Interventions: Device: Active Sentry Handpiece
- Ozil Handpiece: At high IOP settings
  Interventions: Device: Ozil Handpiece

INTERVENTIONS:
Device: Active Sentry Handpiece — With low IOP settings
  Groups: Active Sentry Handpiece
Device: Ozil Handpiece — With high IOP settings.
  Groups: Ozil Handpiece

SUMMARY:
The objective is to assess the efficiency of the Active Sentry handpiece at low intraocular pressure (IOP) compared with the Ozil at high IOP.

DETAILED DESCRIPTION:
This study is a single site, single-masked, randomized, prospective, contralateral eye study of the efficiency of the Active Sentry handpiece at low IOP compared with the Ozil at high IOP.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Be eligible to undergo sequential bilateral uncomplicated cataract surgery.
* Undergo uneventful cataract surgery.
* Gender: Males and Females.
* Both eyes must have same grade of cataract.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Patient under 50 years of age.
* Unable to complete sequential bilateral cataract surgery in both eyes by the same surgeon (JS).
* Patient cataract surgery complicated by posterior capsular tear.
* Any disease state deemed by PI that increases risk of complicated cataract surgery (ie Pseudoexfoliation syndrome, zonular dehiscence, history of eye trauma, RA, prior refractive surgery, etc).

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible test subjects will be 50 years of age or older and who are eligible to undergo sequential bilateral uncomplicated cataract surgery.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Spaulding, DO, Principal Investigator — Cataract and Laser Institute
Locations (1):
- Cataract & Laser Institute, Medford, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Overall (All Participants): Contralateral eye study, flow includes all participants.
  One eye was randomly assigned to either the Active Sentry or Ozil group and the other eye was assigned to the opposite group.
Period: Overall Study
Arm/Group | Overall (All Participants)
Started | 36; 72 eyes
Active Sentry | 36; 36 eyes
Ozil | 36; 36 eyes
Completed | 36; 72 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Groups:
- Overall (All Participants): Contralateral eye study, flow includes all participants
Arm/Group | Overall (All Participants)
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Total Aspiration Time
Time Frame: Day of surgery (Day 0)
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | Active Sentry Handpiece | Ozil Handpiece
Number analyzed (Participants) | 36 | 36
Number analyzed (eyes) | 36 | 36
seconds | 90.1 (16.4) | 85.1 (17.0)

2. Secondary Outcome: Total Fluid Volume
Time Frame: Day of surgery (Day 0)
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: eyes
Arm/Group | Active Sentry Handpiece | Ozil Handpiece
Number analyzed (Participants) | 36 | 36
Number analyzed (eyes) | 36 | 36
mL | 32.8 (4.6) | 33.8 (6.0)

3. Secondary Outcome: Total Phaco Time
Time Frame: Day of surgery (Day 0)
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | Active Sentry Handpiece | Ozil Handpiece
Number analyzed (Participants) | 36 | 36
Number analyzed (eyes) | 36 | 36
seconds | 29.5 (7.3) | 31.0 (7.4)

4. Secondary Outcome: Central Corneal Thickness
Time Frame: 1 week postoperative
Measure: Mean (Standard Deviation); unit: um
Units Other Than Participants: eyes
Arm/Group | Active Sentry Handpiece | Ozil Handpiece
Number analyzed (Participants) | 36 | 36
Number analyzed (eyes) | 36 | 36
um | 554.9 (27.6) | 555.5 (28.8)

5. Other Pre Specified Outcome: Cumulative Dissipated Energy (CDE)
Description: CDE is the amount of ultrasound energy used to remove a cataractous lens. CDE is the power and time of torsional and longitudinal ultrasound delivery modes. It is not expressed in standard units, but is generally unitless. CDE is calculated by the Centurion® Vision System automatically. A lower value is indicative of lower energy used in the eye.
Time Frame: Day of surgery (Day 0)
Measure: Mean (Standard Deviation); unit: unitless
Units Other Than Participants: eyes
Arm/Group | Active Sentry Handpiece | Ozil Handpiece
Number analyzed (Participants) | 36 | 36
Number analyzed (eyes) | 36 | 36
unitless | 5.0 (1.9) | 5.2 (1.7)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Active Sentry Handpiece | Ozil Handpiece
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 1/36 | 2/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Sentry Handpiece (N=36) | Ozil Handpiece (N=36)
corneal edema (Eye disorders) | 0 | 1
iritis (Eye disorders) | 0 | 1
Elevated IOP (Eye disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT05868772/Prot_SAP_000.pdf